CLINICAL TRIAL: NCT00839384
Title: Clinical Study to Evaluate System Safety and Clinical Performance of the AdvisaTM IPG
Brief Title: AdvisaTM IPG Clinical Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: CRDM CE Clinical Department, Medtronic Bakken Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-11

CONDITIONS: Bradycardia; Atrial Tachyarrhythmia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implant Advisa IPG (Experimental): Advisa IPG implant
  Interventions: Device: Advisa IPG

INTERVENTIONS:
Device: Advisa IPG — Implantable Pulse Generator will be implanted

SUMMARY:
The purpose of the Advisa IPG clinical study is to evaluate the overall system safety and clinical performance of the Advisa DR Implantable Pulse Generator (IPG).

DETAILED DESCRIPTION:
The Advisa IPG is an investigational dual chamber pacemaker that provides rate-responsive bradycardia pacing and diagnostics and atrial tachycardia detection and therapy.

The study will be a prospective, non-randomized, multicenter clinical study, conducted.

To allow for sufficient experience with the device, a maximum of 80 subjects may be implanted with the Advisa device. Data will be collected at baseline (enrollment), implant, 1-, 3- and 6- months post implant and every 6 months thereafter or until study closure (whichever occurs first), unscheduled follow-up visits, System Modifications, Technical Observations, Study Deviations, Study Exit, upon notification of new or updated Adverse Events and in case of death.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have an IPG indication for implantation of a dual chamber pacemaker.
* Patients who are geographically stable and available for follow-up at the study center for the duration of the study.
* Patients who have signed a Medical Ethics Committee (MEC) approved Informed Consent form.

Exclusion Criteria:

* Patients with a life expectancy less than the duration of the study.
* Patients with a Class III indication for permanent pacing according to ACC/AHA/NASPE 2002 guidelines.
* Patients with medical conditions that preclude the testing required for all patients by the study protocol or that otherwise limit study participation required for all patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
USADE at 1 month post implant | 1 month
  Confirm safety of the device by assessing the percentage of subjects with an unanticipated serious adverse device effect (USADE) at 1-month post-implant

SECONDARY OUTCOMES:
Advisa IPG system performance | 1 month
  System performance as observed during Holter recordings, Save-to-Disk data and Technical Observations.

CONTACTS AND LOCATIONS:
Overall Officials: Advisa Clinical Study Team, Study Chair — Medtronic Cardiac Rhythm and Heart Failure
Locations (1):
- IKEM, Prague, Czechia